CLINICAL TRIAL: NCT00265291
Title: Antidepressant Treatment of Mexican-Americans: UCLA Pharmacogenetics and Pharmacogenomics Research Group
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Julio Licinio, University of Miami
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: U01GM061394 (NIH)
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-09

CONDITIONS: Major Depressive Disorder; Major Depression; Unipolar Depression
Keywords: Depression; mood disorders; affective disorders; pharmacogenetics; pharmacogenomics
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression; Mood Disorders | interventions — Fluoxetine; Desipramine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluoxetine or desipramine — fluoxetine 5-40 mg/day desipramine 50-150 mg/day
  Other Names: Prozac

SUMMARY:
Our goal is to study pharmacogenetics in Mexican-Americans, using depression treatments as a proof of the concept that pharmacogenetic approaches can be used to optimize treatment strategies for common and complex disorders in this population.

DETAILED DESCRIPTION:
This is a single site, 8-week, double-blinded, placebo lead-in trial with fluoxetine or desipramine. All subjects have a comprehensive psychiatric and medical assessment, and if enrolled, continued with two consecutive phases of the study: 1) A one-week, single-blind placebo lead-in phase to eliminate placebo responders. 2) Subsequent random assignment to one of two treatment groups: fluoxetine 10-40 mg/day or desipramine 50-200 mg/day. Given the proven efficacy of these antidepressant medications, a placebo lead-in period followed by active treatment for all patients has been utilized in order to minimize human subjects at risk.

ELIGIBILITY:
Inclusion Criteria: 1) At least 3 out of 4 grandparents born in Mexico [12]. 2) DSM-IV diagnosis of current, unipolar major depressive episode [13]. 3) 21-Item Hamilton Depression Rating Scale (HAM-D) [14] score of 18 or greater with item #1 (depressed mood) rated 2 or greater. 4) Age between 18-70 years.

-

Exclusion Criteria: 1) Any axis I disorder other than major depressive disorder (e.g. dementia, psychotic illness, bipolar disorder, adjustment disorder) or primary anxiety disorders. 2) Active medical illnesses that could be related to the ongoing depression (e.g. untreated hypothyroidism, recent myocardial infarction or cerebrovascular accident within the past six months, uncontrolled hypertension or diabetes). 3) Current suicidal ideation with a plan and strong intent, or recent serious suicide attempt. 4) Pregnant or lactating women, or women of childbearing age not using contraception. 5) History of electroconvulsive therapy in the last six months. 6) Current use of medications with central nervous system activity which interfere with EEG activity (e.g. benzodiazepines) or any other antidepressant treatment within the 2 weeks prior to enrollment. 7) History of poor response to therapeutic treatment with desipramine or fluoxetine. 8) Illicit drug use and/or alcohol abuse in the last three months. 9) Current enrollment in counseling or psychotherapies.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 1999-11; Primary Completion 2006-05 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The Hamilton Depression Rating Scale (HAM-D) on a weekly basis | 8 weeks

SECONDARY OUTCOMES:
The Hamilton Anxiety Rating Scales (HAM-A), the Global Assessment Scale (GAS), the Beck Depression Inventory (BDI), and the Center for Epidemiological Depression Rating Scale (CES-D) on a weekly basis | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julio Licinio, MD, Principal Investigator — University of Miami
Locations (1):
- Center for Pharmacogenomics, University of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Flores DL, Alvarado I, Wong ML, Licinio J, Flockhart D. Clinical implications of genetic polymorphism of CYP2D6 in Mexican Americans. Ann Intern Med. 2004 Jun 1;140(11):W71. doi: 10.7326/0003-4819-140-11-200406010-00028-w2. No abstract available. PMID 15172931
- [Result] Licinio J, O'Kirwan F, Irizarry K, Merriman B, Thakur S, Jepson R, Lake S, Tantisira KG, Weiss ST, Wong ML. Association of a corticotropin-releasing hormone receptor 1 haplotype and antidepressant treatment response in Mexican-Americans. Mol Psychiatry. 2004 Dec;9(12):1075-82. doi: 10.1038/sj.mp.4001587. PMID 15365580
- [Derived] Wong ML, Arcos-Burgos M, Liu S, Licinio AW, Yu C, Chin EWM, Yao WD, Lu XY, Bornstein SR, Licinio J. Rare Functional Variants Associated with Antidepressant Remission in Mexican-Americans: Short title: Antidepressant remission and pharmacogenetics in Mexican-Americans. J Affect Disord. 2021 Jan 15;279:491-500. doi: 10.1016/j.jad.2020.10.027. Epub 2020 Oct 17. PMID 33128939
- [Derived] Wong ML, Dong C, Flores DL, Ehrhart-Bornstein M, Bornstein S, Arcos-Burgos M, Licinio J. Clinical outcomes and genome-wide association for a brain methylation site in an antidepressant pharmacogenetics study in Mexican Americans. Am J Psychiatry. 2014 Dec 1;171(12):1297-309. doi: 10.1176/appi.ajp.2014.12091165. Epub 2014 Oct 31. PMID 25220861
- [Derived] Licinio J, Dong C, Wong ML. Novel sequence variations in the brain-derived neurotrophic factor gene and association with major depression and antidepressant treatment response. Arch Gen Psychiatry. 2009 May;66(5):488-97. doi: 10.1001/archgenpsychiatry.2009.38. PMID 19414708